CLINICAL TRIAL: NCT01019486
Title: Regadenoson Blood Flow in Type 1 Diabetes (RABIT1D)
Acronym: RABIT1D
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 09-0426
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Results first posted 2015-12-14 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-11

CONDITIONS: Coronary Artery Disease; Type 1 Diabetes Mellitus
Keywords: Myocardial blood flow; Cardiac magnetic resonance imaging; Myocardial perfusion imaging; Coronary artery flow reserve; Regadenoson
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus, Type 1 | interventions — Technetium Tc 99m Sestamibi; regadenoson; gadoteridol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Type 1 Diabetic Subjects (Experimental): Regadenoson 400mcg slow IV bolus to identify assess myocardial blood flow (MBF). Stratified by coronary calcium score of below 100 or greater than score of 100 for low and high risk individuals respectively.
  Interventions: Drug: Regadenoson myocardial perfusion imaging; Drug: Regadenoson MRI myocardial blood flow
- Nondiabetic Subjects (Active Comparator): Regadenoson myocardial perfusion imaging (MPI) Intervention: Regadenoson (400mcg slow IV bolus) stress to assess myocardial blood flow (MBF) and MPI to identify occult coronary artery disease (CAD). These individuals serve as an active control with higher risk non-diabetic individuals with scores greater than 100.
  Interventions: Drug: Regadenoson myocardial perfusion imaging; Drug: Regadenoson MRI myocardial blood flow

INTERVENTIONS:
Drug: Regadenoson myocardial perfusion imaging — Myocardial perfusion imaging at rest and following 400mcg Regadenoson IV bolus pharmacologic stress with 30 mCi of Tc-99m sestamibi injected at both but the studies performed 48 hours apart.
  Other Names: Cardiolite (sestamibi); Regadenoson (Lexiscan)
Drug: Regadenoson MRI myocardial blood flow — CMR assessment of stress myocardial perfusion and blood flow after 400 mcg Regadenoson pharmacologic using gadolinium contrast (gadoteridol) 0.05mmole/kg at stress and rest.
  Other Names: Regadenoson (Lexiscan); Prohance (Gadoteridol)

SUMMARY:
Cardiovascular disease (CVD) remains the major cause of mortality and morbidity in both type 1 (T1D) and type 2 (T2D) diabetes patients; modifications of traditional CVD risk factors have had a limited impact. This project called Regadenoson Blood flow in Type 1 Diabetes (RABIT1D) and is proposed as a sub-study of the Coronary Artery Calcification in Type 1 Diabetes (CACTI) study, which has established a unique cohort of 656 T1D patients (age 20-55, minimal diabetes duration of 10 yrs) and 764 non-diabetic controls. This cohort is being followed for progression of coronary artery calcification (CAC) measured using the electron beam tomography (EBT) for development of clinical CVD. Participants have been well characterized during the baseline examination (4/00-3/02) and two follow-up re-examinations 3 and 6 years later. The study has provided important insights into the risk factors and possible prevention of premature CVD in T1D. We are proposing assess a subset of this population to determine vasodilatory reserve as it relates to early coronary atherosclerosis in T1D.

Hypothesis: that myocardial blood imaging (MBF) reserve can be measured in Type 1 diabetes mellitus (DM) using regadenoson stress cardiac magnetic resonance and that significantly reduced MBF is a marker of extensive atherosclerotic disease correlated to coronary arterial calcification, plaque formation and impaired vasodilatory reserve.

DETAILED DESCRIPTION:
The CACTI cohort is being followed for progression of coronary artery calcification (CAC) for development of clinical CVD and participants have been characterized during the baseline examination (4/00-3/02) and two follow-up re-examinations 3 and 6 years later. We are proposing assess a subset of this population to determine vasodilatory reserve as it relates to early coronary atherosclerosis in T1D. In the CACTI Study sought to determine the relationship between risk factors for CAD and coronary arterial calcification in T1D subjects compared to an age and gender matched control cohort. The trial identified CAC as a high risk marker of CAD and was more extensive in diabetic patients.

T1D patients have more CAC than nondiabetic controls but they also appear to have more impaired coronary vasoreactive function. Impaired response to acetylcholine testing and adenosine vasodilation are reported in diabetic subjects. The relationship between coronary microvascular dysfunction and diabetic cardiomyopathy is supported by observation of similar microvascular abnormalities. Endothelial dysfunction not only precedes and predicts clinical macrovascular disease, but also is an independent prognostic marker of adverse long-term cardiovascular outcomes. Significantly greater CAC in T1D was also noted than in non-DM subjects. There is also a greater rate of increase noted in the CACTI cohort.

Myocardial Flow Reserve by MRI: Myocardial perfusion distribution and myocardial blood flow reserve can be simultaneously assessed using a MRI first-pass Gd contrast injection approach. Rapid MR imaging (MRI) during the first pass injection of Gd compounds is used to assess myocardial perfusion with a spatial resolution of 2-3 mm, and to detect any regional impairments of myocardial blood flow (MBF) that may lead to ischemia. The myocardial perfusion reserve (MPR) is a useful concept for quantifying the vasodilator response. The perfusion reserve can be estimated from the ratio of MBFs during vasodilation and at baseline, similar to that described by labeled microspheres. Assessment of myocardial blood flow and flow reserve by cardiac MR is a robust technique. There is a relationship between CAC and hyperemic flow reserve, although it may be more or less strong depending upon the methodology employed. However, CAC is still a marker of the atherosclerotic process and this process appears to be more aggressive in T1D. The investigation of MBF reserve as a marker of early or more aggressive vasculopathy is important, especially in a disease with significant morbidity and mortality from cardiovascular events.

Regadenoson Vasodilation: Regadenoson is a selective A2A adenosine receptor agonist FDA released as a pharmacologic vasodilator in nuclear stress myocardial perfusion imaging (MPI). It has a higher affinity for A2A receptors than adenosine and is a more potent coronary vasodilator. Adenosine infusion is the gold standard for both invasive and non-invasive assessment of myocardial blood flow reserve, yet regadenoson with potentially greater coronary arterial vasodilation and a simple bolus injection is an ideal agent with which to study differences in CFR between different disease states. Limited data is published on the utility of regadenoson in invasive assessment of CFR and no data are published regarding the utility of this agent in assessing the hyperemic myocardial blood flow response with respect to cardiac MRI.

Research Design and Methods POPULATION CACTI Diabetes Study: We propose to recruit subjects from the CACTI cohort into this sub-study by focusing on individuals completing 6-yr follow-up.

Imaging Studies Non-DM CAC>100 T1D CAC< 100 T1D CAC> 100 MPI 5 10 10 CMR 5 10 10 InvCBF 5 5-10 5-10 Subject will be recruited to complete all three parts of the protocol myocardial perfusion imaging (MPI); cardiac MR assessment of myocardial blood flow reserve (MBF); and only those subject with significant symptoms or clinical indications proceeding to invasive "Catheterization Laboratory" assessment of CBF reserve (Invasive CBF) Aim 1. Determine the relationship between myocardial perfusion index, regional CBF and invasively measured coronary perfusion reserve The first approach will be to assess the differences in myocardial perfusion between T1D and non-DM subjects employing vasodilatory stress with regadenoson. The myocardial perfusion index as described previously will be calculated for each individual. The relative perfusion index will be directly compared to the invasively obtained CBF reserve in each vascular territory assessed.

Stress Myocardial Perfusion Protocols. Subjects will undergo regadenoson stress MPI with 400 mcg administered as a 10 second bolus followed by injection of 30 mCi of Tc-99m-sestamibi. Gated SPECT perfusion imaging is then performed within 30 minutes. A rest study is performed on a separate day with a similar sestamibi dose administered.

Acquisition Protocol. All SPECT studies are performed with parallel hole collimators and gated acquisitions protocol (10% RR window) acquired into 16 time bins. Data Processing of Gated data sets are assessed for mean counts, corrected for dose, decay and time of imaging, are measured in each segment utilizing 4D-MSPECT (INVIA, Ann Arbor, Michigan). MPI is defined as the corrected stress counts divided by corrected rest counts.

Statistical Analysis: Based upon our prior experience approximately a third of the T1D subjects will have a MP index of less that 1.5 to direct compare to the invasive measured flow reserve. This maybe treated as a binary variable or as a continuous variable by combining all T1D subject compared to the non-DM control subjects. Data will be analyzed using unpaired t-test, linear and logistic regression. Continuous variables are expressed as mean ± standard deviation (SD) and are compared across groups by use of unpaired t-tests. All statistical analysis will be performed using two-sided tests with p < 0.05 considered statistically significant.

Aim 2. Measure coronary blood flow using Regadenoson stress CMR to determine the MBF reserve in type 1 DM subjects compared to non-diabetic controls. Using the method of a two compartment model with K trans function analysis, we will determine the myocardial blood flow reserve by cardiac MR. This approach will use regadenoson bolus as the vasodilator for the hyperemic response of the coronary arterial bed. We will assess the relationship of MBF reserve or lack of reserve to disease state i.e T1D to non-DM subjects. In addition we will regionally compare MBF reserve to the MP index obtained from radionuclide techniques by coronary vascular territories. Similarly CAC values obtained at the 6-yr CACTI follow-up study will be directly compared to blood flow measurement within coronary vascular distributions.

CMR Protocol: An IV injection into the antecubital vein and connected to a power injector will be performed in the MR scanner for functional and perfusion imaging (Symphony 1.5 T, Siemens Medical). All images are acquired with a 4 channel phased array surface coil. Blood flow imaging is performed in three short-axis simultaneous slices (basal, mid and apical) acquired during an initial bolus injection of gadolinium (0.04 mmol/kg at a rate of 5 ml/sec) followed by a 10-ml saline flush administered using the power injector. ProHance is used due to its lower viscosity as the contrast agent. The short-axis slices are acquired using a SSFP imaging sequence with, TR/TE/flip 185ms/1.2ms/50 degrees dynamically acquired and inserted into a 330x 380 matrix). Images are acquired using a field of view ranging from 280 to 400 mm. A first perfusion scan will be performed at rest, followed by a second scan during maximal vasodilation about 15 min later. Hyperemia will be initiated with administration of 400 mcg bolus injection of regadenoson and acquisition started 1 minute post regadenoson administration. Subjects will be monitored using MRI compatible blood pressure monitoring and single lead ECG monitoring.

Data analysis Quantitative analysis of the MR blood flow data will be performed on a Leonardo Workstation using Argus perfusion analysis software. Images were registered manually by adjusting the horizontal and vertical registration of each frame. The left and right ventricular blood pool and six myocardial regions will be analyzed to extract the linear slope during the initial signal increase as well as the starting and peak signal intensities. To extract the slope, base, and peak signals, a line was manually fitted to the upslope signal (typically 4-6 time points), and the base and peak positions of the upslope data were manually identified. Normalized slope (SlopeN) was calculated by division by the left ventricular blood pool slope, and the net signal gain (SG) determined by subtracting the initial from the peak signal intensity. The myocardial flow reserve index was calculated for each myocardial region as the ratio of the normalized hyperemic time-intensity slope to the normalized baseline time-intensity slope.

Statistical Analysis: Based upon prior experience in the literature approximately a third of the T1D subjects will have a MP index of less than 1.5 to direct compare to the invasive measured flow reserve. Data will be analyzed using unpaired t-test, linear and logistic regression.

Aim 3. Determine the relationship between CBF reserve in vascular distributions to the degree of coronary arterial calcification.

Coronary artery calcification. All returning patients have previously undergone EBT scan. These data as described above will be used to compare to the new MPI, CMR myocardial blood flow reserve, and to the invasively measured CFR. Regional change will determined within standard coronary vascular distributions.

Flow Reserve Substudy Protocol: High-risk diabetics with CAC> 100 (n=10) and stratified random sample high risk non-diabetics (n=10) will be studied. The inclusion of subjects with an abnormal perfusion reserve is important, because this value identified subjects with high risk in the first phase of the study and therefore is used to select individuals with high risk of cardiac events that clinically would undergo invasive assessment of coronary anatomy. Perfusion imaging will then be the test that stratifies subjects into an additional higher risk than the CAC > 100. Selected patients identified as part of Specific Aim 2 will undergo a clinically indicated cardiac catheterization and baseline CFR study. Coronary angiography is the clinically accepted standard for evaluation and diagnosis of coronary artery disease.

Subsequently, coronary artery vasodilator reserve will be assessed using the regadenoson intravenous challenge technique measured as the coronary flow reserve and fraction flow reserve assess by a Doppler flow guide wire.

Methods for Flow Reserve:Selective coronary angiography is performed using standard technique with 5F diagnostic catheters in the LCA and RCA. The artery or interest determined by the abnormal area of myocardial perfusion by SPECT or MR imaging will be interrogated. The artery of interest will be cannulated with a 6F or 7F Guide catheter. A 0.014 in x 300cm pressure and Doppler-tipped guidewire (CombMap XT, Volcano Corp) will be advanced into the distal bed of the vessel of interest. After optimization of the pressure and Doppler signal, velocity and pressure measurements will be obtained at rest and after induction of maximal hyperemia with an intravenous bolus of regadenoson. Coronary flow reserve (CFR) will be measured in the target vessel of interest after 1-2 minutes following the IV bolus. Absolute CFVR will be calculated as the ratio of hyperemic to baseline average peak flow velocity and the relative CFVR as the ratio of the absolute CFVR in the target vessel to the absolute CFVR in the reference artery. FFR and CFR values will be categorized according to published cut-off values of 0.75 and 2.0, respectively.

ELIGIBILITY:
Inclusion Criteria:

* 1. Inclusion Criteria Nondiabetic controls High-risk (n=5)

  1. Completed visit 6yr f/u CACTI Trial
  2. No history of previous MI, revascularization or angina
  3. CAC > 100
  4. Stratified random sample to reflect age-sex- distribution of the high risk diabetic group T1Diabetic subjects High-risk group (n= 10)

  <!-- -->

  1. Completed visit 6yr f/u CACTI Trial
  2. No history of previous MI, revascularization or angina
  3. CAC > 100
  4. preferably MPR of > 1.5 T1Diabetic subjects Lower-risk group (n= 10)

  <!-- -->

  1. Completed visit 1.A and 1.B CACTI Trial
  2. No history of previous MI, revascularization or angina
  3. CAC < 100

     Exclusion Criteria:

  2. Exclusion Criteria:
  1. Pregnant or lactating women, women who plan to become pregnant
  2. Claustrophobia
  3. Moderate or severe congestive heart failure at baseline, Left ventricular ejection fraction (LVEF) < 25%
  4. Uncontrolled hypertension
  5. Unwillingness to complete all components of the study
  6. Significant CAD or prior revascularization
  7. Smoker
  8. Subject cannot have >50% reduction in lumen diameter of left main coronary artery
  9. Asthma requiring daily bronchodilators
  10. Methylxanthine therapy
  11. Moderate to severe renal insufficiency: GFR < 40 mL/min

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert A. Quaife, M.D, Principal Investigator — University of Colorado, Denver
Locations (4):
- United States (4):
  - Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
  - University of Colorado Denver, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - University Hospital, the University of Colorado Health Sciences Center, Denver, Colorado

REFERENCES:
- [Background] Mekkaoui C, Jadbabaie F, Dione DP, Meoli DF, Purushothaman K, Belardinelli L, Sinusas AJ. Effects of adenosine and a selective A2A adenosine receptor agonist on hemodynamic and thallium-201 and technetium-99m-sestaMIBI biodistribution and kinetics. JACC Cardiovasc Imaging. 2009 Oct;2(10):1198-208. doi: 10.1016/j.jcmg.2009.06.013. PMID 19833310
- [Background] Tomillero A, Moral MA. Gateways to clinical trials. Methods Find Exp Clin Pharmacol. 2009 Jul-Aug;31(6):397-417. PMID 19798455
- [Background] Mahmarian JJ, Cerqueira MD, Iskandrian AE, Bateman TM, Thomas GS, Hendel RC, Moye LA, Olmsted AW. Regadenoson induces comparable left ventricular perfusion defects as adenosine: a quantitative analysis from the ADVANCE MPI 2 trial. JACC Cardiovasc Imaging. 2009 Aug;2(8):959-68. doi: 10.1016/j.jcmg.2009.04.011. PMID 19679284
- [Background] Hage FG, Heo J, Franks B, Belardinelli L, Blackburn B, Wang W, Iskandrian AE. Differences in heart rate response to adenosine and regadenoson in patients with and without diabetes mellitus. Am Heart J. 2009 Apr;157(4):771-6. doi: 10.1016/j.ahj.2009.01.011. Epub 2009 Mar 6. PMID 19332209
- [Background] Libby P, Nathan DM, Abraham K, Brunzell JD, Fradkin JE, Haffner SM, Hsueh W, Rewers M, Roberts BT, Savage PJ, Skarlatos S, Wassef M, Rabadan-Diehl C; National Heart, Lung, and Blood Institute; National Institute of Diabetes and Digestive and Kidney Diseases Working Group on Cardiovascular Complications of Type 1 Diabetes Mellitus. Report of the National Heart, Lung, and Blood Institute-National Institute of Diabetes and Digestive and Kidney Diseases Working Group on Cardiovascular Complications of Type 1 Diabetes Mellitus. Circulation. 2005 Jun 28;111(25):3489-93. doi: 10.1161/CIRCULATIONAHA.104.529651. No abstract available. PMID 15983263

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began 7-22-2010 and ended 12-30-2011. We recruited from subjects of the Coronary Artery Calcification in Type 1 (CACTI) Diabetes Study (R01HL61753) included type 1 diabetic patients (duration, diabetes 10 yrs) and non-diabetic controls (spouses or friends of these diabetic patients, focusing on individuals completing 6-yr follow-up..
Pre-assignment Details: Twenty-five subjects planned with 26 consented with one excluded with significant renal disease. A total of 25 myocardial perfusion imaging studies; 23 MRI myocardial blood flow (MBF) MRI studies performed of which 23 yielded analyzable. A total of 3 subject meet criteria to proceed to invasive coronary flow reserve measurements
Groups:
- Non Diabetic Controls: Subjects with Coronary Artery Calcium (CAC score> 100 in the CACTI Stdy)
- Type 1 Diabetes Low Risk Group: Subjects with T1DM for at least 10 years and CAC < 100
- Type 1 Diabetes High Risk Group: Subjects with T1DM for at least 10 years and CAC > or = 100
Period: Overall Study
Arm/Group | Non Diabetic Controls | Type 1 Diabetes Low Risk Group | Type 1 Diabetes High Risk Group
Started | 5 | 5 | 16
Completed | 4 | 4 | 15
Not Completed | 1 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: mean age value with standard deviation.
Groups:
- Total: Total of all reporting groups
Arm/Group | Non Diabetic Controls | Type 1 Diabetes Low Risk Group | Type 1 Diabetes High Risk Group | Total
Number analyzed (Participants) | 4 | 4 | 15 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 13 | 21
  >=65 years | 0 | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (1.6) | 59.3 (10.1) | 57.3 (5.2) | 59.8 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 4 | 5
  Male | 3 | 4 | 11 | 18
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 15 | 23

OUTCOME MEASURES:

1. Primary Outcome: Coronary Blood Flow Assessment With Regadenoson Stress by Cardiac MRI Between Non-diabetic and Type 1 Diabetic Subjects.
Description: Measurement of Myocardial blood flow measurements (MBF) and myocardial perfusion index obtained from 6 regions within the mid ventricular LV short axis slice.
Time Frame: 1 month
Population: Determine the MBF obtained from cardiac MRI from 6 regions of the mid-ventricular LV myocardium and a ratio between stress/rest myocardial blood flow ratio. Differences between group were compared using a unpaired "t" test analyzed for: control(Con) vs T1DM low risk; Con. vs T1DM High Risk; and T1DM low vs high risk.
Measure: Mean (Standard Deviation); unit: percentage of StressMBF/ Rest MBF
Arm/Group | Non Diabetic Controls | Type 1 Diabetes Low Risk Group | Type 1 Diabetes High Risk Group
Number analyzed (Participants) | 4 | 4 | 15
percentage of StressMBF/ Rest MBF | 2.19 (0.3) | 1.81 (0.6) | 1.95 (0.7)
Statistical Analysis 1: Comparison: Non Diabetic Controls vs Type 1 Diabetes Low Risk Group; Independent Student t test between arms with two tailed analysis; Test type: Superiority or Other; p < 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: Non Diabetic Controls vs Type 1 Diabetes High Risk Group; Independent Student t test between arms with two tailed analysis; Test type: Superiority or Other; p < 0.05, t-test, 2 sided
Statistical Analysis 3: Comparison: Type 1 Diabetes Low Risk Group vs Type 1 Diabetes High Risk Group; Independent Student t test between groups with two-tailed analysis; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

2. Secondary Outcome: Measured Coronary Blood Flow is Directly Correlated With Coronary Flow Reserve Measured Invasively in the Cardiac Catheterization Laboratory After Regadenoson Pharmacologic Stress.
Description: Regional coronary blood flow reserve (CFR) in a target artery (defined on MPI study) compared to flow in a less diseased atherosclerotic vessel following vasodilator response to intravenously administered regadenoson.
Time Frame: within 6 months
Population: Only 3 individuals met the prescribed perfusion defect on MPI study to proceed to the CFR measurement arm of the study. Therefore numbers were too small for statistical comparison and only mean value and standard deviation of the flow ratio(CFR measurements) are reported..
Measure: Mean (Standard Deviation); unit: CFR ratio
Groups:
- Abnormal MPI Study: These subjects demonstrated abnormal radionuclide myocardial perfusion imaging studies with perfusion defects in response to regadenoson stress. The perfusion defect qualified the subject to participated in invasive CFR measurements. Coronary arteries within the region of the perfusion defect were cannulated for CFR measurements. Flow measurements were performed in the 2 normal vessels and the abnormal vessel both at rest and following regadenoson administration to calculated CFR values..
Arm/Group | Abnormal MPI Study
Number analyzed (Participants) | 3
CFR ratio | 1.5 (0.5)
Statistical Analysis 1: Comparison: Abnormal MPI Study; No analysis was performed due to limited data; Test type: Non-Inferiority or Equivalence — If sufficient subjects were enrolled then it would be expected that the MRI measurement of myocardial blood flow MBF would similar or equivalent to the invasively measured CFR in response to intravenous regadenoson administration; p = 0.05, Wilcoxon (Mann-Whitney); None insufficient data = 2.0

3. Secondary Outcome: Myocardial Perfusion Index
Description: Myocardial perfusion indices radionuclide stress and rest images and were obtained from 6 regions within the mid ventricular LV short axis slice. Each was corrected for decay and standardized to a 30 mCi administered dose for each part of a two day study.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: percentage of Ratio Stress/ rest counts
Arm/Group | Non Diabetic Controls | Type 1 Diabetes Low Risk Group | Type 1 Diabetes High Risk Group
Number analyzed (Participants) | 4 | 4 | 15
percentage of Ratio Stress/ rest counts | 1.09 (.19) | 1.4 (.60) | 1.12 (.32)
Statistical Analysis 1: Comparison: Non Diabetic Controls vs Type 1 Diabetes Low Risk Group vs Type 1 Diabetes High Risk Group; Comparison between groups using a two-tailed Student t test; Test type: Superiority or Other; p < .05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Event were recorded over the 18 months of the study.
Arm/Group | Non Diabetic Controls | Type 1 Diabetes Low Risk Group | Type 1 Diabetes High Risk Group
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5 | 0/16
Other Adverse Events (participants affected / at risk) | 0/4 | 0/5 | 0/16

LIMITATIONS AND CAVEATS:
3 subject had visual perfusion defects, leading to a small % of individuals being referred for invasive CFR measurements. MBF values were less than reported, either from microvascular disease in T1D subjects or the order of rest first then stress.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No